CLINICAL TRIAL: NCT03042702
Title: A Phase 2 Study of Kevetrin (Thioureidobutyronitrile) in Subjects With Platinum-Resistant/Refractory Ovarian Cancer
Brief Title: A Phase 2 Study of Kevetrin in Subjects With Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovation Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTIX-KEV-201
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Results first posted 2018-12-27 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Cohort Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Kevetrin 250 mg/m2 IV Cohort 1 (Experimental): Kevetrin 250 mg/m2 IV per dose every other day (q.o.d.)/ 3 doses per week (750 mg/m2 per week), for 3 weeks (single cycle; total 9 doses) Follow-up For 3 weeks after Kevetrin treatment ends
  Interventions: Drug: Kevetrin
- Kevetrin 350 mg/m2 IV Cohort 2 (Experimental): Kevetrin 350 mg/m2 IV per dose every other day (q.o.d.)/ 3 doses per week (1050 mg/m2 per week), for 3 weeks (single cycle; total 9 doses) Follow-up For 3 weeks after Kevetrin treatment ends
  Interventions: Drug: Kevetrin

INTERVENTIONS:
Drug: Kevetrin — Kevetrin dose to associated cohort
  Other Names: Cohort
  Arms: Kevetrin 250 mg/m2 IV Cohort 1
Drug: Kevetrin — Kevetrin dose to associated cohort
  Arms: Kevetrin 350 mg/m2 IV Cohort 2

SUMMARY:
Cellceutix has developed Kevetrin (thioureidobutyronitrile), belonging to an anti-proliferative p53 activator pharmacological class, for the treatment of cancer. Nonclinical studies have demonstrated that Kevetrin induces apoptosis by activation of wild type p53 and induces apoptosis in mutant p53 cells by degradation of oncogenic mutant p53.

In this Phase 2 study, two different short-term treatment regimens of Kevetrin will be evaluated for safety, tolerability, changes in biomarkers/objective tumor response, and to evaluate the pharmacokinetics of Kevetrin when administered to subjects with platinum-resistant/refractory ovarian cancer.

DETAILED DESCRIPTION:
This is an open label, dose-escalation trial to study the safety, biomarker changes (including modulation of p53), objective tumor response changes, and pharmacokinetics following administration of two different treatment regimens of Kevetrin over a 3-week period to subjects with platinum-resistant/refractory ovarian cancer. Following the 3 weeks of Kevetrin dosing, subjects are to be followed up for 3 weeks after completion of Kevetrin treatment. Standard of care treatment, as medically appropriate and per local guidelines, outside of this study protocol can commence after the collection of the post-Kevetrin treatment biomarker samples (collected on Day 21±1 day). The patient population recruited into this study includes those ovarian cancer patients that have platinum resistant/refractory disease, defined as disease progression/relapse within 6 months following the last administered dose of platinum therapy (resistant), or lack of response or disease progression while receiving the most recent platinum based therapy (refractory), respectively. Patients may or may not have had additional treatment (e.g., Doxil) prior to entry in this study.

A total of approximately 10 study participants are planned to be enrolled in two cohorts of approximately 5 subjects per cohort, with enrollment in a sequential, dose-escalating fashion. Investigators and subjects will be aware of the treatment cohort into which they are recruiting. Cohort details and the planned doses are:

Cohort 1 (n=5) Kevetrin Cycle - Kevetrin 250 mg/m2 IV per dose every other day (q.o.d.)/ 3 doses per week (750 mg/m2 per week), for 3 weeks (single cycle; total 9 doses); Follow-up for 3 weeks after Kevetrin treatment ends Cohort 2 (n=5) Kevetrin Cycle - Kevetrin 350 mg/m2 IV per dose every other day (q.o.d.)/ 3 doses per week (1050 mg/m2 per week), for 3 weeks (single cycle; total 9 doses); Follow-up for 3 weeks after Kevetrin treatment ends Cohorts 1 and 2 will be conducted in a sequential fashion, with safety data from cohort 1 evaluated by an independent Data Monitoring Committee (DMC). The DMC will make appropriate recommendations based on the available safety data as regards the intent of progressing to the higher dose cohort 2.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated written informed consent to participate in the clinical study
2. Non-pregnant female adults at least 18 years of age at time of informed consent
3. Histologically confirmed serous epithelial ovarian cancer with peritoneal metastases
4. Platinum resistant/refractory disease, defined as disease progression/relapse within 6 months following the last administered dose of platinum therapy (resistant), or lack of response or disease progression while receiving the most recent platinum based therapy (refractory), respectively
5. Measurable disease, as determined by radiologist evaluator, with at least 1 unidimensional measurable lesion (target lesion) by RECIST v.1.1 that has not previously been irradiated or biopsied
6. Presence of non-target lesions that have not previously been irradiated or biopsied; to allow for collection of needle-biopsies at Screening and after completion of Kevetrin treatment
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. Adequate hematologic and organ function as confirmed by laboratory values at Screening:

   1. Bone marrow function: Absolute neutrophil count (ANC) ≥ 1500 Cells/μL (with no evidence that this ANC was induced or supported by granulocyte colony stimulating factors)
   2. Hemoglobin ≥ 9 g/dL (with no RBC transfusions within 7 days of Screening)
   3. Platelets ≥ 100,000 cells/μL (with no evidence that this platelet count was induced or supported by a platelet-stimulating agent)
   4. Renal function: creatinine ≤ 1.5 x ULN
   5. Hepatic function: total bilirubin ≤ 1.5 x ULN; ALT and AST ≤ 3 x ULN; alkaline phosphatase ≤ 2.5 x ULN
   6. Neurologic function: neuropathy (sensory and motor) ≤ CTCAE Grade 1
   7. Coagulation status: prothrombin time (PT) ≤ 1.5 ULN or INR within normal limits; and partial thromboplastin time (PTT) ≤ 1.2 × ULN
9. Women of child-bearing potential are required to use effective contraception throughout the study period. Effective contraception methods include:

   1. Total abstinence (if this is the usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. (Subject must agree to use contraception should they become sexually active while on the study.)
   2. Surgical sterilization (hysterectomy and/or bilateral oophorectomy) or tubal ligation at least six weeks before start of study treatment.
   3. Male partner sterilization, occurring at least 6 months prior to screening. For female subjects on the study, the vasectomized male partner should be their sole partner.
   4. Double barrier method: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.
   5. Oral*/ injected/ implanted/ transdermal hormonal contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), e.g., hormone vaginal ring.
   6. Intrauterine device or intrauterine system. *Stable oral contraception use (on the same pill) for a minimum of 3 months before taking study treatment.

   Women are considered post-menopausal and not of child-bearing potential if they have had 12 consecutive months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical hysterectomy and/or bilateral oophorectomy or tubal ligation at least six weeks ago.
10. Estimated life expectancy of at least 6 months, in the Investigator's opinion
11. Willing and able to comply with scheduled visits, study assessments and laboratory tests, and other study procedures

Exclusion Criteria:

1. Unwilling to allow removal of tumor biological samples for analysis, i.e., biopsies of tumor lesions, and/or collection of ascites fluid from abdominal ascites (if present)
2. Non epithelial tumor, including malignant mixed Müllerian tumors without high grade serous component, or ovarian tumors with low malignant potential (i.e., borderline tumors)
3. Known presence of central nervous system metastases
4. Presence of tumor metastases causing significant pleural disease/effusion unilaterally or bilaterally (significant pleural effusion is defined by need for thoracentesis more frequently than once every 21 days)
5. Presence of ascites that requires paracentesis more frequently than once every 21 days.
6. A history of another primary cancer that has been active or treated within the past 3 years prior to start of study treatment, with the exception of adequately treated/resected: basal cell or squamous cell skin carcinoma or actinic keratoses; or carcinoma in situ of the breast or of the cervix; or non-invasive malignant colon polyps
7. Persistent toxic effects with severity of CTCAE grade 2 or greater (excluding alopecia) caused by previous treatment
8. History of arterial or deep venous thromboembolism within the 12 months prior to enrollment
9. Clinically significant cardiac disease, including:

   1. Myocardial infarction or unstable angina < 6 months prior to enrollment
   2. New York Heart Association (NYHA) Grade II or greater congestive heart failure
   3. Cardiac arrhythmia requiring medication (does not include asymptomatic atrial fibrillation with controlled ventricular rate)
10. Electrocardiogram (ECG) obtained at Screening which shows QTc prolongation or other medically relevant abnormalities which may affect subject safety or interpretation of study results
11. At a higher than average risk, in the Investigator's opinion, of bowel perforation (e.g., symptoms of partial or complete bowel obstruction, recent (within 6 months) history of fistula or bowel perforation, requirement for total parenteral nutrition and continuous hydration)
12. Active or chronic recurrent systemic infections that require continuous antimicrobial therapy during the Kevetrin study period
13. Past medical history of infection with HIV, hepatitis B or hepatitis C
14. Ongoing or recent history of any other uncontrolled and/or clinically significant systemic disease or condition which, in the Investigator's medical opinion, should exclude participation in the study
15. Less than 3 weeks between major surgery and planned start of study treatment; major incisions must have healed
16. Less than 4 weeks since last treatment for ovarian cancer
17. Any investigational or experimental therapy or procedure or participation in any interventional trial within 4 weeks or 5 half-lives (whichever is longer) prior to start of study treatment
18. Women of child-bearing potential who are pregnant or nursing (lactating)
19. Previous participation in a clinical study of Kevetrin
20. History of alcohol or substance abuse, unless in full remission for more than 6 months prior to start of study treatment
21. Any other severe acute or chronic medical or psychiatric condition or test abnormality(ies) that, in the Investigator's opinion, puts the subject at significant risk, could confound the study results, or may interfere significantly with the subject's participation in the study

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 2 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Bertolino, MD, Study Director — Cellceutix Corporation
Locations (2):
- United States (2):
  - Cancer Research, Lebanon, New Hampshire
  - Cancer Research, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled in the "Kevetrin 350 mg/m2 IV"/"Cohort 2" Arm/Group.
Groups:
- Kevetrin 250 mg/m2 IV/Cohort 1: Kevetrin 250 mg/m2 IV per dose every other day (q.o.d.)/ 3 doses per week (750 mg/m2 per week), for 3 weeks (single cycle; total 9 doses) Follow-up For 3 weeks after Kevetrin treatment ends
  Kevetrin: Kevetrin dose to associated cohort
Period: Overall Study
Arm/Group | Kevetrin 250 mg/m2 IV/Cohort 1
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Kevetrin 250 mg/m2 IV/Cohort 1
Number analyzed (Participants) | 2
Age, Customized [Count of Participants; unit: Participants]
  54 years old | 1
  71 years old | 1
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Reporting of Adverse Events, and severity of adverse events
Time Frame: 6 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Kevetrin 250 mg/m2 IV/Cohort 1
Number analyzed (Participants) | 2
Participants
  TEAE Yes | 2
  TEAE No | 0

2. Primary Outcome: Number of Participants With Changes in Biomarkers
Description: Changes in RNA and/or protein level of pre-specified biomarkers associated with the p53 signalling pathway and apoptosis will be compared between pre-treatment sample (tumor biopsy, ascites fluid, and peripheral blood) and post-treatment sample (tumor biopsy, ascites fluid, and peripheral blood)
Time Frame: 3 Weeks
Population: All
Measure: Count of Participants; unit: Participants
Arm/Group | Kevetrin 250 mg/m2 IV/Cohort 1
Number analyzed (Participants) | 2
Participants
  Observed biomarker changes | 2
  No observed biomarker changes | 0

3. Secondary Outcome: Number of Participants by RECIST Tumor Response Category
Description: Number of subjects in each response category (complete response, partial response, stable disease or progressive disease) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
  CR (Complete Response): Disappearance of all target lesions PR (Partial Response) : At least a 30% decrease in the sum of the longest diameters of target lesions PD (Progressive Disease) : At least a 20% increase in the sum of the longest diameters of target lesions SD (Stable Disease) : Small changes that do not meet above criteria
Time Frame: 3 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Kevetrin 250 mg/m2 IV Cohort 1
Number analyzed (Participants) | 2
Participants
  Complete response | 0
  Stable disease | 2
  Partial response | 0
  Progressive disease | 0

4. Secondary Outcome: Maximum Plasma Concentration of Kevetrin (Cmax) on Days 1 and 5
Description: Measurement of Kevetrin systemic concentrations from collected blood samples. Due to low number of subjects individual values are presented.
Time Frame: Prior to dosing, During 3h infusion: 60(±5) min, 120(±5) min, and 2 min prior to end of infusion, i.e., 178 min. Post infusion: 0.5 hour (±5 min), 1 hour (±5 min), 2 hour (±5 min), 4 hour (±10 mins), 6 hour (±30 mins) [optional], and 24(±4) hour
Measure: Number; unit: ng/mL
Arm/Group | Kevetrin 250 mg/m2 IV Cohort 1
Number analyzed (Participants) | 2
ng/mL
  Subject 002-001 Cmax Day 1 | 1820
  Subject 002-001 Cmax Day 5 | 1840
  Subject 002-002 Cmax Day 1 | 2410
  Subject 002-002 Cmax Day 5 | 2450

5. Secondary Outcome: Time to Reach the Maximum Plasma Concentration of Kevetrin (Tmax) on Days 1 and 5
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Number; unit: hours
Arm/Group | Kevetrin 250 mg/m2 IV Cohort 1
Number analyzed (Participants) | 2
hours
  Subject 002-001 Tmax Day 1 | 2.97
  Subject 002-001 Tmax Day 5 | 2.97
  Subject 002-002 Tmax Day 1 | 2.97
  Subject 002-002 Tmax Day 5 | 1.97

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUCt) on Days 1 and 5
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Number; unit: hours*ng/mL
Arm/Group | Kevetrin 250 mg/m2 IV Cohort 1
Number analyzed (Participants) | 2
hours*ng/mL
  Subject 002-001 AUCt Day 1 | 6851
  Subject 002-001 AUCt Day 5 | 6531
  Subject 002-002 AUCt Day 1 | 8141
  Subject 002-002 AUCt Day 5 | 8385

ADVERSE EVENTS:
Time Frame: AEs were collected from Screening thru End of Study. approximately 6 weeks
Groups:
- Cohort 1: Kevetrin 250 mg/m2 IV per dose every other day (q.o.d.)/ 3 doses per week (750 mg/m2 per week), for 3 weeks (single cycle; total 9 doses) Follow-up For 3 weeks after Kevetrin treatment ends
  Kevetrin: Kevetrin dose to associated cohort
Arm/Group | Cohort 1
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=2)
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Fatigue (Gastrointestinal disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT03042702/Prot_SAP_000.pdf